CLINICAL TRIAL: NCT02178254
Title: A Randomized, Safety, Tolerability and Pharmacokinetics 3-Period Crossover Study Comparing 2 Single Doses of ZTI-01 and Monurol® in Healthy Subjects
Brief Title: Safety, Tolerability and PK 3-Period Crossover Study Comparing 2 Single Doses of ZTI-01 and Monurol® in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 13-0064; HHSN272201500005I
Record Dates: First submitted 2014-06-26; First posted 2014-06-30 (Estimated); Last update posted 2016-04-04 (Estimated); Status verified 2015-01

CONDITIONS: Pseudomonas Infection
Keywords: Pseudomonas aeruginosa, ZTI-101, phosphonic acid derivative, Monurol, fosfomycin tromethamine
MeSH Terms: conditions — Pseudomonas Infections | interventions — Fosfomycin

ARMS (3):
- Sequence 3 (Experimental): N=10 subjects receive 3grams oral sachet of Monurol in Period 1; 1.0gram of Intravenous (IV) ZTI-01 for Period 2 (1-hour infusion); and 8.0 grams IV ZTI-01 for Period 3.
  Interventions: Drug: Fosfomycin tromethamine; Drug: Fosfomycin disodium
- Sequence 1 (Experimental): N=10 subjects receive 1.0gram of Intravenous (IV) ZTI-01 for Period 1 (1-hour infusion); 8.0 grams IV ZTI-01 for Period 2 (1-hour infusion); and 3grams oral sachet of Monurol in Period 3.
  Interventions: Drug: Fosfomycin tromethamine; Drug: Fosfomycin disodium
- Sequence 2 (Experimental): N=10 subjects receive 8.0 grams IV ZTI-01 for Period 1(1-hour infusion); 3grams oral sachet of Monurol in Period 2 and 1.0gram of IV ZTI-01 for Period 3 (1-hour infusion)
  Interventions: Drug: Fosfomycin tromethamine; Drug: Fosfomycin disodium

INTERVENTIONS:
Drug: Fosfomycin tromethamine — A phosphonic acid derivative is the mono-acid salt of Fosfomycin with Tromethamine. Sequence 1-3 receive 3 grams oral sachet
Drug: Fosfomycin disodium — ZTI-01 is a phosphonic acid derivative formulated as a disodium salt intravenous formulation. ZTI-01 acts by inhibiting peptidoglycan assembly, thereby disrupting cell wall synthesis. Sequence 1-3 receive 1 gram and 8 grams of Intravenous ZTI-01 for 1-hour infusion

SUMMARY:
The objective is to determine the safety, tolerability and pharmacokinetics (PK) of 2 single doses of ZTI-01 (1g and 8g infused over 1-hr) and a single dose of the Reference Label Drug, Monurol® (oral sachet, 3g). Subjects will be randomized to a treatment sequence prior to dosing on Day 1 of Period 1 prior to study screening.

DETAILED DESCRIPTION:
This is a Phase 1 single-dose, randomized, 3-Period, crossover study conducted at a single center. A total of 30 healthy subjects, aged 18-45years, will be randomized to receive one of 3 treatment sequences. The duration of study will be approximately 18-26 days and subject participation will be the duration of study. Each treatment sequence will be enrolled in parallel and each subject will receive all 3 treatments in crossover fashion. Each subject will complete Screening, Baseline, and Treatment Phases. The Screening Phase will be conducted on an outpatient basis within 35 days of admission (Day -1 of Period 1). All subjects admitted to the study center the day before dosing in each treatment period (Day -1; check-in) for pre-dosing assessments and will remain in the study center through 48 hours post-dose for each Period. Final baseline qualification will only be evaluated prior to randomization for Treatment Period 1. Each one of the periods will be separated by a 3 (minimum) to 7 days (maximum) washout period. The Treatment Phase will be comprised of 3 crossover periods (duration Day-1 to 48 hours post dose). Each crossover period will include a single dose of study drug under fasting conditions followed by post-dose safety assessments and blood and urine collection for PK measures through 48 hours post-dose; each period will be separated by a 3 to 7 days washout. Subjects will remain in the study center for all 3- study treatment periods (Day -1 to 48 hours post dosing) and will be discharged after the 48-hour sampling timepoint (if safety parameters are acceptable to the Investigator on Day 3).

ELIGIBILITY:
Inclusion Criteria:

To be considered for study enrollment, subjects must meet all of the inclusion criteria:

* Healthy men and women from 18 to 45 years of age with no clinically significant findings on medical history, physical examination, vital signs, 12-lead electrocardiogram (ECG) or clinical laboratory evaluation that were performed at Screening and Day -1.
* Body Mass Index (BMI) between 18-30 kg/m^2, inclusive; and a total body weight > 50 kg (110 lbs).
* Post-menopausal women with amenorrhea for at least 2 years with an FSH in the post-menopausal range as well as surgically sterile women (documented history of oophorectomy and/or hysterectomy, tubal ligation or tubal occlusion) will be eligible.
* Females of childbearing potential must use an acceptable birth control method (e.g., condom plus spermicide, combined oral contraceptive, implant, injectable, indwelling intrauterine device, sexual abstinence, or a vasectomized partner) throughout the study and for 4 weeks following initiation of dosing with study drug.
* Male subjects must either had a vasectomy or agree to use a double barrier method of contraception, condom plus spermicide (or diaphragm plus spermicide in female partner) from the time of dosing with the study drug in Period 1 through 4 weeks following initiation of dosing with study drug.
* Nicotine-free by history (cigarettes, pipe, cigar, chewing tobacco, nicotine patch) for at least 30 days before Day -1 and urine cotinine at pre-study screening and Day -1 <400 ng/mL).
* Able to abstain from grapefruit, grapefruit juice, grapefruit-containing products or alcoholic beverages within 48 hours before Day -1 and throughout the inpatient period.
* Willing to remain in the study facility and agree to abide to the Quintiles Phase 1 Unit House Rules for the duration of the inpatient study period.
* Have a high probability for compliance and completion of the study.
* Sign a dated, witnessed, written informed consent form

Exclusion Criteria:

Subjects must meet none of the following study criteria at Study Day -1, Period 1:

* History or presence of any psychiatric or emotional disorder that might prevent the successful completion of the study.
* Any surgical or medical condition that in the opinion of the investigator could interfere with drug absorption, distribution, metabolism, or excretion or any condition that may place the subject at increased risk while participating in the study. Examples of the conditions for exclusion: previous bariatric surgery, cardiovascular disease, renal impairment, renal disease, liver disease, chronic pulmonary disease, venous insufficiency, peripheral edema, borderline hypertension systolic pressure over > 140mmHg and or diastolic pressure >90 mmHg, serum sodium or liver enzymes above the upper limit, Regarding the last two conditions, one repeat is allowed at both screening and check-in to determine eligibility.
* Any history or presence of clinically significant allergic conditions (e.g., recurrent dermatitis or drug hypersensitivity reactions).
* Have cancer or have a history of cancer (with exceptions of a few types of cancer, e.g. recent removal of basal cell skin carcinoma) within the past five years.
* Irritable bowel syndrome or any gastrointestinal disease (including frequent nausea due to migraine) within 30 days prior to study day 1, Period 1.
* History or presence of lactose intolerance.
* History of alcohol abuse within 12 months of study day 1, Period 1.
* History of intolerance or hypersensitivity to phosphonic acid derivative antibiotics or any of its constituents
* Use of any prescription drugs within 30 days of administration of the study drug
* Involvement in other investigational studies of any type (drugs, devices, procedures) within 30 days of screening.
* Blood or blood products donation within 60 days of Day -1.
* Use of any non-prescription medications, vitamins, licorice (in large amounts) or dietary supplements within 7 days of administration of the study drug. Excluded from this list is intermittent use of acetaminophen at doses of </=2 g/day. Herbal supplements must be discontinued 7 days prior to the initial dose of study drug.
* Consumption of more than 300 mg of caffeine per day (>3 cups of coffee or 6-12 ounces of soda) within 7 days prior to dosing.
* Presence of any acute illness within 7 days of Day -1 in any Study Period.
* Breastfeeding or a positive serum pregnancy test at the Screening Visit or on Day -1 in any Study Period
* Positive tests for human immunodeficiency virus (HIV 1 and 2) antibodies, hepatitis B surface antigen (HBsAg) and/or hepatitis C (HCV) antibody.
* Positive urine drug or alcohol screen at the Screening Visit or on Day -1
* Weight loss or gain of > 10 percent within 30 days of Day -1.
* Females whose hemoglobin is <11.8 g/dL or males whose hemoglobin is <13.8g/dL.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-08; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics: Maximum measured plasma concentration (Cmax), area under the concentration versus time curve (AUC0-t and AUC0-inf), time to peak concentration (tmax), terminal elimination half-life (t1/2), terminal-phase elimination rate constant). | Study periods 1, 2 and 3, Day 1 through Day 3
Pharmacokinetics: Volume of distribution (Vd) or apparent volume of distribution (Vd/F) as appropriate, clearance (CL) or apparent Clearance (CL/F) as appropriate, renal Clearance (CLr) and Fraction Bioavailable as appropriate | Study periods 1, 2 and 3, Day 1 through Day 3
Adverse events (AEs) will be monitored and recorded | Study periods 1, 2 and 3, screening through Day 3, including washout periods
Assessed safety and tolerability via physical examinations, vital signs, standard 12-lead electrocardiograms, and clinical laboratory tests | Study periods 1, 2 and 3, screening through Day 3

CONTACTS AND LOCATIONS:
Locations (1):
- Quintiles Phase I Services - Overland Park, Overland Park, Kansas, United States